CLINICAL TRIAL: NCT01999465
Title: Neuromuscular Electrical Stimulation (NMES) Efficacy on Patients With Neonatal Brachial Plexus Palsy (NBPP)
Brief Title: NMES Efficacy on Patients With NBPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Spring Arbor University (Unknown)
Responsible Party: Principal Investigator, Lynda Yang, MD, PhD, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MedSAU-NMES
Record Dates: First submitted 2013-10-29; First posted 2013-12-03 (Estimated); Results first posted 2018-12-14 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Neonatal Brachial Plexus Palsy
Keywords: Brachial plexus injury; Brachial plexus palsy; Neonate
MeSH Terms: conditions — Neonatal Brachial Plexus Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard NMES cohort (Active Comparator): Patients who will apply standard NMES device.
  Interventions: Device: Standard NMES device
- Sham NMES cohort (Sham Comparator): Patients who will apply sham NMES device.
  Interventions: Device: Sham NMES device

INTERVENTIONS:
Device: Standard NMES device — Blinded parents will follow the NMES parent instructions and place the NMES on the biceps muscle of their child for 30 minutes every day for three months.
  * Rate(35 Hz)
  * Width (300 us)
  * Ch1 Ramp+ (2 seconds)
  * On Time 1 (10 seconds)
  * Ch1 Ramp - (2 seconds)
  Other Names: Neuromuscular electrical stimulation (NMES)
  Arms: Standard NMES cohort
Device: Sham NMES device — Blinded parents will follow the NMES parent instructions and place the NMES on the biceps muscle of their child for 30 minutes every day for three months.
  * Rate(35 Hz)
  * Width (48 us)
  * Ch1 Ramp+ (0 seconds)
  * On Time 1 (0 seconds)
  * Ch1 Ramp - (0 seconds)
  Arms: Sham NMES cohort

SUMMARY:
Neonatal Brachial Plexus Palsy (NBPP), characterized by weakness and sensory loss in the affected arm, results from damage in the prenatal period to the nerves extending from the spine to the arm. Proper stretching and exercise of the joints and affected arm from the time of diagnosis can greatly assist in the development of healthy movement of the limb. Additionally, neuromuscular electrical stimulation has been shown to be an effective treatment in other neural disorders and therefore its effectiveness in NBPP is worth studying.

In the case of NBPP patients, the loss in normal arm function can be observed very early. Young patients will often neglect using the affected arm or modify motions to avoid the use of the biceps muscle, specifically in hand to mouth actions such as gripping a bottle or placing toys or other objects in the mouth. A goal of this study is to test the effectiveness of NMES on improving the biceps muscle Medical Research Council (MRC) strength and active range of motion (AROM).

The subjects of this study are newborns between the ages of 3-9 months who are already a part of the University of Michigan Brachial Plexus program. Parents of the children will be trained to perform the neuromuscular electrical stimulation therapy at home using the EMPI Continuum unit for 30 minutes each day and monthly follow up appointments will be performed be the research occupational therapists throughout three month study period.

Parents of the participants will complete a questionnaire before and during the study period to help analyze for confounders and gather data regarding parent compliance and NMES effectiveness. To detect the effectiveness of NMES, two cohort groups using standard units and sham units will be recruited and compare with data analysis.

The investigators predict that the NMES will effectively improve the ability of the neonate to increase use of the affected arm, specifically in muscle strength biceps MRC score and AROM.

DETAILED DESCRIPTION:
The purpose of this study is to investigate whether the use of Neuromuscular Electrical Stimulation (NMES), via the Empi® Continuum unit, will improve the ability with which children with Neonatal Brachial Plexus Palsy (NBPP) are able to use their biceps muscle in activities of daily living. We will examine the British Medical Research Council (MRC) muscle strength and participants' ability to perform active range of motion (AROM) movements. Patients will be divided into two groups with one group receiving NMES and the other receiving sham NMES. We plan to analyze the effects of this one treatment intervention of NMES to determine if the device improves the function of the biceps muscle strength and motion.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 3-9 months at time of enrollment
* NBPP patients who receive care from University Of Michigan Brachial Plexus Palsy clinic
* All gender/race/financial backgrounds
* active range of motion (AROM) elbow flexion <150°
* All Narakas grades
* British Medical Research Council (MRC) grade 2- or 4 for biceps brachii

Exclusion Criteria:

* Brachial Plexus patients require needing surgical repair
* Patients with any existing secondary medical conditions
* Patients with elbow contracture greater than 5°
* British Medical Research Council (MRC) grade 5 for biceps brachii
* active range of motion (AROM) elbow flexion =150°
* Non-English speaking families
* Children already using NMES unit

Ages: 3 Months to 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Yang, MD, PhD, Principal Investigator — Neurosurgery Department, University of Michigan Health System
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard NMES Cohort: Patients who will apply standard NMES device.
  Standard NMES device: Blinded parents will follow the NMES parent instructions and place the NMES on the biceps muscle of their child for 30 minutes every day for three months.
  * Rate(35 Hz)
  * Width (300 us)
  * Ch1 Ramp+ (2 seconds)
  * On Time 1 (10 seconds)
  * Ch1 Ramp - (2 seconds)
- Sham NMES Cohort: Patients who will apply sham NMES device.
  Sham NMES device: Blinded parents will follow the NMES parent instructions and place the NMES on the biceps muscle of their child for 30 minutes every day for three months.
  * Rate(35 Hz)
  * Width (48 us)
  * Ch1 Ramp+ (0 seconds)
  * On Time 1 (0 seconds)
  * Ch1 Ramp - (0 seconds)
Period: Overall Study
Arm/Group | Standard NMES Cohort | Sham NMES Cohort
Started | 10 | 10
Completed | 10 | 7
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard NMES Cohort | Sham NMES Cohort | Total
Number analyzed (Participants) | 10 | 7 | 17
Age, Continuous [Mean (Standard Deviation); unit: months] — age is described as months
  months | 4 (2) | 4 (1) | 4 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 9 | 5 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 7 | 17
NBPP-involved side [Count of Participants; unit: Participants]
  Left | 5 | 2 | 7
  Right | 5 | 5 | 10
Narakas [Count of Participants; unit: Participants] — Narakas grade is determined by a single surgeon via either: 1) physical examination and neurological assessment at approximately 1 week of age or at initial clinical appointment, or 2) mother's or obstetrician's report of child's arm/hand movements at birth. The Narakas grade is grouped into Grade I-II versus III-IV in the current study.
  Narakas Groups I and II are considered to be less extensive NBPP injury and Groups III and IV are more extensive NBPP injury.
  Participants
    Narakas I-II | 8 | 5 | 13
    Narakas III-IV | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Upper Extremity Muscle Strength
Description: One of the two-blinded occupational therapists will conduct the evaluation at enrollment and 3-month follow-up clinic visit. In this study, we will evaluate the biceps strength using the British Medical Research Council (MRC) grading system. The British Medical Research Council (MRC) grading system for muscle strength is based on a scale from 0 (minimum score, not testable), 1, 2, 3, 4, to 5 (maximum score, normal strength); higher score means better outcome. British Medical Research Council (MRC) grade 2 or higher is functional in terms of muscle power. In current study, we will examine the change of biceps British Medical Research Council (MRC) grade from baseline to 3-month.
Time Frame: Baseline to 3-month.
Population: One in the Standard NMES cohort was lost of follow-up and two in the sham cohort were lost of follow-up at 3 months.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Standard NMES Cohort | Sham NMES Cohort
Number analyzed (Participants) | 9 | 5
score on a scale | 1 [0 to 5] | 1 [0 to 5]
Statistical Analysis 1: Comparison: Standard NMES Cohort vs Sham NMES Cohort; Test type: Other; p = 0.40, Wilcoxon (Mann-Whitney); We applied Wilcoxon-Mann Whitney test with the Null hypothesis that there is no difference between 2 arms

2. Primary Outcome: Change From Baseline in Upper Extremity Range of Motion
Description: One of the two-blinded occupational therapists will assess the active range of motion (AROM) of elbow flexion using goniometer at enrollment and 3-month follow-up clinic visit. The minimum degree is 0 and the maximum degree is 150; the higher degree means better outcome. We will then examine the change of elbow flexion active range of motion (AROM) from baseline to 3-month.
Time Frame: Baseline to 3-month.
Population: One in the Standard NMES cohort was lost of follow-up and two in the sham cohort were lost of follow-up at 3 months.
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Standard NMES Cohort | Sham NMES Cohort
Number analyzed (Participants) | 9 | 5
degree | 55 (38) | 29 (25)
Statistical Analysis 1: Comparison: Standard NMES Cohort vs Sham NMES Cohort; Test type: Other; p = 0.20, t-test, 2 sided

3. Other Pre Specified Outcome: Change From Baseline in Spontaneous Hand-to-Mouth Movement
Description: Study coordinators will conduct one-minute video recording with patient in supported sitting position in a chair or seated on parents lap at initial and monthly clinic visits. A toy, pacifier, or bottle will be provided to trigger patient's spontaneous hand-to-mouth movement. The frequency of hand to mouth motion will be recorded and separated out as to the positioning of the elbow. We are evaluating the motion to determine if the motion of the elbow flexion is against gravity, (the arm held at the side of the body or in an adducted position) or in gravity-eliminated position, (the arm held away from the body or in an abducted position). We are looking at the strength of the biceps in its ability to lift the arm against gravity during functional hand to mouth activities. The NMES unit will not be in use during the videotaping process; we are looking at the spontaneous movement of the extremity.
Time Frame: Baseline to 3-month.
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Change From Baseline in Participant's Current Therapy
Description: Parents will complete a survey asking participant's current therapy program, including therapy type, setting, frequency, duration, other treatment activities, splint usage, home range of motion exercise program and its frequency and duration at initial and monthly follow-up visits. The purpose of this survey is to help us understand whether there are potential confounders that could affect the study result.
Time Frame: Baseline to 3-month.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Standard NMES Cohort | Sham NMES Cohort
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 0/10 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT01999465/Prot_SAP_000.pdf